CLINICAL TRIAL: NCT01427907
Title: Randomized,Multi-center,Phase IV, 2-arm,Open-Label,Cross-over Study to Demonstrate the Equivalence of Calcium Acetate Oral Solution and Sevelamer Carbonate Tablets in Hemodialysis Patients
Brief Title: Equivalence of Calcium Acetate Oral Solution and Sevelamer Carbonate Tablets in Hemodialysis Patients
Acronym: COS-002
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COS-002
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Kidney Disease
Keywords: Serum phosphorus levels
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — calcium acetate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phoslyra - Calcium Acetate Oral Solution (Experimental): The investigational compound is calcium acetate oral solution (COS) or Phoslyra. It is a pale, light greenish-yellow clear liquid with a characteristic black cherry odor and flavor for oral ingestion. Each 5 mL of COS contains 667 mg calcium acetate equal to 169 mg of elemental calcium. Each subject will follow their usual prescription.COS will be taken either prior to or during meals and snacks.
  Interventions: Drug: Calcium acetate oral solution (COS)
- Sevelamer Carbonate (Active Comparator): Sevelamer carbonate is an anion exchange resin that binds phosphate in the gastrointestinal tract and is a buffered form of sevelamer hydrochloride developed for the treatment of hyperphosphatemia in End-Stage Renal Disease (ESRD) patients. Each film-coated tablet of sevelamer carbonate (trade name Renvela™) contains 800 mg of sevelamer carbonate on an anhydrous basis. Subjects will receive sevelamer tablets according to their prescription.
  Interventions: Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: Calcium acetate oral solution (COS) — Each subject will undergo two separate treatment periods. Subjects will ingest either COS or sevelamer for 28 days (Treatment Period 1) and then switch to the other binder for 28 days (Treatment Period 2).
  Other Names: Phoslyra
  Arms: Phoslyra - Calcium Acetate Oral Solution
Drug: Sevelamer carbonate — Each subject will undergo two separate treatment periods. Subjects will ingest either COS or sevelamer for 28 days (Treatment Period 1) and then switch to the other binder for 28 days (Treatment Period 2).
  Other Names: Renvela
  Arms: Sevelamer Carbonate

SUMMARY:
The purpose of this study is to demonstrate equivalence of calcium acetate oral solution and sevelamer carbonate in maintaining serum phosphorus levels

This is a phase IV, multicenter, randomized, open-label, cross-over study to assess the equivalence of a liquid formulation of a calcium-based phosphate binder, COS, to sevelamer carbonate tablets, in hemodialysis dependent Chronic Kidney Disease subjects (CKD). The aim of the study is to maintain serum phosphorus level and establish equivalence between COS and sevelamer carbonate tablets.

DETAILED DESCRIPTION:
Total 40 subjects will be randomized for participation into the study The subjects are Hemo-dialysis Dependent Chronic Kidney Disease (CKD) Stage 5D patients who are able to give informed consent to the study, and taking the phosphate binder sevelamer carbonate tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age able to give written informed consent to the study
* Hemodialysis dependent chronic kidney disease stage 5D patients
* Taking sevelamer carbonate tablets or sevelamer hydrochloride as phosphate binder monotherapy
* Taking 3 or more sevelamer carbonate or sevelamer hydrochloride tablets per day

Exclusion Criteria:

* Estimated life expectancy of less than 6 months and for cancer patients, an Eastern Cooperative Oncology Group (ECOG) Performance Status >1
* Active malignancy within the past 5 years. Basal or squamous cell skin cancer is not exclusionary. History of malignancy is not an exclusion
* Known hypersensitivity reaction to calcium-based phosphate binders
* Anticipated renal transplantation during the study
* Pregnant or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Katanko, MD, Principal Investigator — Renal Research Institute
Locations (4):
- United States (4):
  - St. Raphael's Dialysis Center, New Haven, Connecticut
  - North Haven Dialysis, North Haven, Connecticut
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dialysis Clinic (UMDC), New York, New York

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 subjects signed the informed consent form (ICF), 5 subjects were not eligible, and 1 eligible subject withdrew the ICF prior to randomization.
Groups:
- Sequence I: COS (4 Weeks) Then Sevelamar (4 Weeks): Patient receive Calcium Acetate Oral Solution (COS) for 4 weeks then cross over to Sevelamer tablets for 4 weeks.
- Sequence II: Sevelamer (4 Weeks) Then COS (4 Weeks): Patient receive Sevelamer tablets for 4 weeks, then cross over to take COS for 4 weeks.
Period: Overall Study
Arm/Group | Sequence I: COS (4 Weeks) Then Sevelamar (4 Weeks) | Sequence II: Sevelamer (4 Weeks) Then COS (4 Weeks)
Started | 20 (Randomized) | 18 (Randomized)
Completed | 17 (Completed study) | 14 (Completed study)
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sequence I: COS Then Sevelamer: Sequence I: Calcium Acetate Oral Solution for 4 weeks then Sevelamer Carbonate for 4 weeks
- Sequence II: Sevelamer Then COS: Sevelamer Carbonate for 4 weeks then Calcium Acetate Oral Solution for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Sequence I: COS Then Sevelamer | Sequence II: Sevelamer Then COS | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (16.3) | 57 (20.2) | 59 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 15 | 9 | 24
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Serum Phosphorus Levels
Description: The average phosphorus level of non-missing laboratory assessments from the last two weeks of each treatment period for each subject
Time Frame: 2 weeks
Population: Modified intent-to-treat: subjects who were randomized, received at least one prescribed dose of the study medication and provided at least one of the last 4 laboratory assessments of each treatment period
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Calcium Acetate Oral Solution: Calcium Acetate Oral Solution for periods 1 and 2
- Sevelamer Carbonate: Sevelamer Carbonate for periods 1 and 2
Arm/Group | Calcium Acetate Oral Solution | Sevelamer Carbonate
Number analyzed (Participants) | 32 | 32
mg/dL | 4.6 (1.20) | 4.6 (0.93)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Calcium Acetate Oral Solution: Sequence I: Calcium Acetate Oral Solution for periods 1 and 2
Arm/Group | Calcium Acetate Oral Solution | Sevelamer Carbonate
Serious Adverse Events (participants affected / at risk) | 2/38 | 1/38
Other Adverse Events (participants affected / at risk) | 13/38 | 6/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Acetate Oral Solution (N=38) | Sevelamer Carbonate (N=38)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — due to cellulitis to both legs
Bacteremia; cellulitis, fever (Infections and infestations) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Acetate Oral Solution (N=38) | Sevelamer Carbonate (N=38)
hematemesis (Renal and urinary disorders) | 1 (1) | 0 (0)
squamous cell carcinoma removed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
hypercalcimia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
left uper quadrant discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
arm pain (General disorders) | 0 (0) | 1 (1)
sharp stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
strong acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Last Patient Last Visit (LPLV) was on 06-July-2012 and last site close out visit was 31 May 2013. Due to inadvertent study deviations, no reliable conclusions can be drawn from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No